CLINICAL TRIAL: NCT00025441
Title: MMT 98 Study For Metastatic Disease Rhabdomyosarcoma And Other Malignant Soft Tissue Sarcoma Of Childhood
Brief Title: Combination Chemotherapy in Treating Children With Metastatic Rhabdomyosarcoma or Other Malignant Mesenchymal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Collaborators: Children's Cancer and Leukaemia Group (Other); Societe Francaise Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068961; SIOP-MMT-98; SFOP-SIOP-MMT-98; CCLG-SIOP-MMT-98; EU-20126; STS-1998
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-11

CONDITIONS: Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: chondrosarcoma; small intestine leiomyosarcoma; fibrosarcomatous osteosarcoma; embryonal childhood rhabdomyosarcoma; alveolar childhood rhabdomyosarcoma; pleomorphic childhood rhabdomyosarcoma; mixed childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; extraosseous Ewing sarcoma/peripheral primitive neuroectodermal tumor; childhood fibrosarcoma; childhood synovial sarcoma; childhood malignant hemangiopericytoma; childhood liposarcoma; childhood alveolar soft-part sarcoma; childhood leiomyosarcoma; childhood angiosarcoma; childhood epithelioid sarcoma; childhood malignant mesenchymoma; stage IV uterine sarcoma; uterine leiomyosarcoma; ovarian sarcoma; previously untreated childhood rhabdomyosarcoma; childhood desmoplastic small round cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma; Chondrosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Fibrosarcoma; Hemangiopericytoma, Malignant; Liposarcoma; Hemangiosarcoma; Malignant mesenchymal tumor; Desmoplastic Small Round Cell Tumor | interventions — Dactinomycin; Filgrastim; Carboplatin; Cyclophosphamide; Doxorubicin; Epirubicin; Etoposide; Ifosfamide; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children with metastatic rhabdomyosarcoma or other malignant mesenchymal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival of children with metastatic rhabdomyosarcoma or other malignant mesenchymal tumors treated with one of two different chemotherapy regimens based upon risk group.
* Determine the role of low-intensity maintenance chemotherapy after intensive conventional chemotherapy in standard-risk children.
* Determine the value of a therapeutic window in high-risk children.
* Determine the role of sequential high-dose chemotherapy with peripheral blood stem cell transplantation in achieving complete response in high-risk children.
* Determine the complete response, overall survival, and event-free survival in high-risk children.

OUTLINE: This is a multicenter study. Patients are stratified according to risk group (standard vs high).

Standard-risk patients:

* Initial chemotherapy: Patients receive vincristine IV on day 1 for weeks 1-7. Patients also receive dactinomycin IV on day 1 and ifosfamide IV over 1 hour on days 1-3 of week 1. Patients then receive carboplatin IV over 1 hour and epirubicin IV over 6 hours on day 1 of week 4. Patients then receive ifosfamide IV over 1 hour and etoposide IV over 4 hours on days 1-3 of week 7. Treatment repeats every 8 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. After the second course, patients with less than 50% partial response (PR) are removed from study.

Patients with parameningeal disease undergo radiotherapy 5 days a week for about 8 weeks beginning at week 9.

* Maintenance chemotherapy: Patients receive cyclophosphamide IV over 1 hour, vincristine IV, and dactinomycin IV on day 1. Treatment repeats every 3 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.

Patients who remain in PR at week 17 undergo radiotherapy for about 9 weeks beginning at week 18.

High-risk patients:

* Initial chemotherapy: Patients receive window study drug carboplatin IV over 1 hour or doxorubicin on day 1. Treatment repeats every 3 weeks for 2 courses.

Patients receive high-dose cyclophosphamide IV over 1 hour on days 1-3 of week 7. Beginning on day 8, patients receive filgrastim (G-CSF) IV or subcutaneously (SC) daily until day 13. Patients may undergo peripheral blood stem cell (PBSC) collection.

Patients receive high-dose etoposide IV over 24 hours on days 15-17. Beginning on day 22, patients receive G-CSF IV or SC daily until day 27.

Patients receive high-dose cyclophosphamide IV over 1 hour on days 29-31. Beginning on day 36, patients receive G-CSF IV or SC daily until day 42. Patients may undergo PBSC collection if not previously performed. Patients who achieve complete response (CR) are removed from study.

Patients receive high-dose carboplatin IV over 1 hour on days 44-48. Patients undergo PBSC reinfusion on day 52. Beginning on day 55, patients receive G-CSF IV or SC daily until blood counts recover.

* Maintenance chemotherapy: Patients receive maintenance chemotherapy comprising cyclophosphamide, vincristine, and dactinomycin in the same manner as the standard-risk patients.

Patients with parameningeal disease and those not achieving CR undergo radiotherapy beginning at week 17. Patients achieving CR, unless metastatic disease is resected, undergo radiotherapy beginning on week 15.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 8-30 standard-risk patients will be accrued for this study within 4 years. A total of 15-75 high-risk patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic rhabdomyosarcoma or other malignant mesenchymal tumors

  * Standard risk defined as:

    * Less than 10 years of age
    * No bone or bone marrow involvement
  * High risk defined as:

    * At least 10 years of age OR
    * Bone or bone marrow involvement
* Diagnosed less than 8 weeks ago
* Previously untreated disease except for initial surgery within the past 8 weeks

PATIENT CHARACTERISTICS:

Age:

* 6 months to under 18 years

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* Concurrent radiotherapy allowed

Surgery:

* See Disease Characteristics

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-11; Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather P. McDowell, MD, Study Chair — Royal Liverpool Children's Hospital, Alder Hey; Annabel B.M. Foot, Study Chair — Bristol Royal Hospital for Children; Christophe Bergeron, Study Chair — Centre Leon Berard
Locations (22):
- Centre Leon Berard, Lyon, France
- Our Lady's Hospital for Sick Children, Crumlin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Leeds Cancer Centre at St. James's University Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland

REFERENCES:
- [Result] McDowell HP, Foot AB, Ellershaw C, Machin D, Giraud C, Bergeron C. Outcomes in paediatric metastatic rhabdomyosarcoma: results of The International Society of Paediatric Oncology (SIOP) study MMT-98. Eur J Cancer. 2010 Jun;46(9):1588-95. doi: 10.1016/j.ejca.2010.02.051. Epub 2010 Mar 24. PMID 20338746